CLINICAL TRIAL: NCT01471665
Title: A Randomised, Double-blind, Placebo-controlled, Cross-over Study to Evaluate the Effect of Treatment With Repeat Dose GSK2190915 as an add-on to Current Therapy on the Percentage of Neutrophils in Induced Sputum in Asthmatic Patients With Elevated Sputum Neutrophils
Brief Title: GSK2190915 Neutrophilic Asthma Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 115134
Record Dates: First submitted 2011-08-18; First posted 2011-11-16 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — 3-(3-tert-butylsulfanyl-1-(4-(6-ethoxypyridin-3-yl)benzyl)-5-(5-methylpyridin-2-ylmethoxy)-1H-indol-2-yl)-2,2-dimethylpropionic acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- GSK2190915 100mg (Experimental): This is a crossover study so patients will receive 100mg of GSK2190915 once daily for up to 16 days followed by a wash out period of at least 14 days before they cross over onto the placebo arm of the study.
  Interventions: Drug: GSK2190915 100mg
- Placebo (Placebo Comparator): This is a crossover study so patients will receive placebo once daily for up to 16 days followed by a wash out period of at least 14 days before they cross over onto the GSK2190915 100mg arm of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2190915 100mg — GSK2190915 is a high affinity 5-lipoxygenase-activating protein (FLAP) inhibitor. Dosing will occur once daily for up to 16 days.
  Arms: GSK2190915 100mg
Drug: Placebo — Placebo will be administered once daily for up to 16 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect on repeat doses of GSK2190915 in asthmatic patients with a high percentage of neutrophils in their sputum. GSK2190915 will be given as an add on to current therapy, and its effects on the percentage of sputum neutrophils in the patients will be assessed.

DETAILED DESCRIPTION:
This is a randomised, double blind, placebo-controlled, two-way cross-over study to evaluate the effect of treatment with repeat dose GSK2190915, a 5-lipoxygenase-activating protein (FLAP) inhibitor, as an add-on to current therapy on the percentage of neutrophils in induced sputum in asthmatic patients with elevated sputum neutrophils. Approximately 20 subjects will be enrolled onto the study to ensure that approximately 14 evaluable subjects complete the study. All subjects will receive oral placebo and GSK2190915 100mg once daily for up to 16 days. Sputum neutrophilia will be assessed prior to treatment and on treatment. Key assessments: sputum cell counts, biomarker samples in sputum, blood and urine, and pharmacokinetics. Safety will be assessed by vital signs, electrocardiograms (ECGs), clinical laboratory safety tests and collection of adverse events (AEs).

GSK2190915 is a high affinity 5-lipoxygenase-activating protein (FLAP) inhibitor that attenuates the production of leukotrienes, through the blockage of the first committed step in the leukotriene pathway, 5-lipoxygenase (5-LO) activation. Leukotrienes are potent inflammatory molecules produced mainly by mast cells, eosinophils, monocytes/macrophage and neutrophils in response to allergic or inflammatory stimuli. As GSK2190915 reproducibly inhibits the production of leukotriene B4 (LTB4) and cysteinyl leukotrienes (cysLTs) both in vitro and in vivo it has strong potential utility in the treatment of asthma.

ELIGIBILITY:
Inclusion Criteria:

* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) < 2xUpper limit of normal (ULN); alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Males and females ages 18 years old and above.
* An established clinical history of asthma in accordance with the definition by the GINA Guidelines.
* Subjects who are stable on their current treatment for at least one month prior to first dose and for the duration of the study.
* Persistent sputum neutrophilia in the absence of infection. Persistent is defined at being met at Screening and Visit 1 of Treatment Period 1. At least one sputum sample must show neutrophils ≥ 50%. The other sample must be > 45%.
* A female subject is eligible to participate if she is of:

  * Non-childbearing potential defined as pre-menopausal females with a documented (medical report verification) hysterectomy or double oophorectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum Follicle Stimulating Hormone (FSH) levels > 40 mIU/mL and estradiol < 40 pg/ml (<140 pmol/L) or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods specified in the protocol if they wish to continue their Hormone Replacement Therapy (HRT) during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
  * Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow up visit, or at least 6 days after last dose.
* Signed and dated written informed consent is obtained from the subject
* The subject is able to understand and comply with the protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* The subject has tested positive for Human Immunodeficiency Virus ev1(HIV) antibodies.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Past or present disease, which as judged by the investigator or medical monitor, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, gastrointestinal disease, hepatic disease, renal disease, haematological disease, neurological disease, endocrine disease or pulmonary disease (excluding asthma but including but not confined to chronic bronchitis, emphysema, bronchiectasis, eosinophilic bronchitis or pulmonary fibrosis).
* History of asthma exacerbations or acute intercurrent respiratory illness (viral respiratory syndrome, bronchitis, pneumonia) for a four week period before the screening visit.
* History of life-threatening asthma, defined as an asthma episode that required intubations and/or was associated with hypercapnia, respiratory arrest and/or hypoxic seizures.
* FEV1 < 1 litre post salbutamol.
* Clinically significant abnormalities in vital signs or safety laboratory analysis at screening.
* The subject has a clinically significant QT duration corrected for heart rate (QTc) value at screening.
* The subject has a positive pre-study urine drug or urine or breath alcohol screen. A minimum list of drugs that will be screened for include Amphetamines, Barbiturates, Cocaine, Opiates, Cannabinoids and Benzodiazepines.
* Administration of injectable steroids within 6 weeks of screening.
* Administration of any vaccinations within 2 weeks of screening or during the study.
* Administration of biological therapies within 3 months of the screening visit or during the study.
* Subject is undergoing allergen desensitisation therapy.
* Administration of OATP1B1 substrates from 2 weeks before dosing, and until all follow up assessments are completed.
* Subject is unable to abstain from taking prescription or non-prescription drugs (including vitamins and dietary or herbal supplements) including non-steroidal antiinflammatory drugs (NSAIDs), anti-depressant drugs, anti-histamines and antiasthma, anti-rhinitis or hay fever medication, with the exception of ICS, Long Acting Beta Agonist (LABA), montelukast and short action beta agonists, within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication until completion of the follow-up visit, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study.
* The subject has participated in a study with a new molecular entity during the previous 3 months or has participated in 4 or more clinical studies in the previous 12 months prior to the first dosing day.
* History of blood donation (500 mL) within 3 months of starting the clinical study.
* History of alcohol abuse or the subject regularly drinks more than 28 units of alcohol in a week if male, or 21 units per week if female. One unit of alcohol is defined as a medium (125 ml) glass of wine, half a pint (250 ml) of beer or one measure (25 ml) of spirits.
* There is a risk of non-compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The numbers of neutrophils in induced sputum in asthmatic subjects (average of absolute and percentage count on Visit 4 and Visit 5) | 13 - 16 days post treatment with 100mg GSK2190915 or placebo once daily
  Pharmacodynamics

SECONDARY OUTCOMES:
The levels of LTE4 in urine, LTB4-glucuronide in urine and LTB4 in sputum supernatant in asthmatic subjects | Over 13 - 16 days post treatment with 100mg GSK2190915 or placebo once daily
  Pharmacodynamics
The levels of high sensitive C-reactive protein (hsCRP) and other biomarkers (for example IL-17) in blood in asthmatic subjects | Over 13 - 16 days post treatment with 100mg GSK2190915 or placebo once daily
  Pharmacodynamics
Changes in symptoms in asthmatic subjects compared to placebo using the asthma control questionnaire | Over 13 - 16 days post treatment with 100mg GSK2190915 or placebo once daily
  Safety and tolerability and efficacy
Changes in lung function as measured by Forced Expiratory Volume in one second (FEV1) in subjects with asthma | Over 13 - 16 days post treatment with 100mg GSK2190915 or placebo once daily
  Safety and tolerability and efficacy
Plasma concentrations of GSK2190915 following repeated doses in asthmatic subjects | On days 13 - 16 days post treatment with 100mg GSK2190915 or placebo once daily
  Pharmacokinetics
Incidence of treatment emergent adverse events in asthmatic subjects and vital signs, electrocardiograms and safety laboratory parameters in asthmatic subjects | Over 13 - 16 days post treatment with 100mg GSK2190915 or placebo once daily
  Safety and tolerability and effiacy
The levels of biomarkers in sputum supernatant, for example IL-17, IL-8, neutrophil elastase and myeloperoxidase, as samples permit, in asthmatic subjects | Over 13 - 16 days post treatment with 100mg GSK2190915 or placebo once daily
  Pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Glasgow, Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Chaudhuri R, Norris V, Kelly K, Zhu CQ, Ambery C, Lafferty J, Cameron E, Thomson NC. Effects of a FLAP inhibitor, GSK2190915, in asthmatics with high sputum neutrophils. Pulm Pharmacol Ther. 2014 Feb;27(1):62-9. doi: 10.1016/j.pupt.2013.11.007. Epub 2013 Dec 10. PMID 24333186
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 115134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register